CLINICAL TRIAL: NCT06738589
Title: The Inflate Study; Defining the Soft Palate in the Upper Airway Flow Pathway
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Collaborators: The University of Auckland (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: U1111-1315-8696
Record Dates: First submitted 2024-12-02; First posted 2024-12-17 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Focus of the Study is the Anatomy of the Soft Palate; Non-invasive Ventilation
Keywords: Soft Palate; MRI; NIV; Airway
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MRI without positive pressure therapy (No Intervention): Healthy volunteers having their upper airway scanned with MRI without the addition of positive airway pressure therapy (NIV)
- MRI with positive pressure (Experimental): Healthy volunteers having their upper airway scanned with MRI with the addition of positive airway pressure therapy (NIV)
  Interventions: Device: non-invasive ventilation

INTERVENTIONS:
Device: non-invasive ventilation — Non-invasive ventilation adds positive pressure to the upper airway via a mask on the face.
  Arms: MRI with positive pressure

SUMMARY:
The goal of this clinical trial is to understand the impact of the size and shape of the soft palate on gas airflow in the upper airway in healthy volunteers. Utilizing Magnetic Resonance Imaging (MRI), this study aims to investigate:

* How does soft palate anatomy change in different body positions?
* What is the impact of positive pressure therapy, in the form of non-invasive ventilation (NIV) on soft palate anatomy? Researchers will compare MRI data without positive pressure to with positive pressure imaging to see if the addition of positive pressure impacts the size and shape of the soft palate.

Researchers will also utilize measures of upper airway resistance to assess the impact of soft palate anatomy of airflow dynamics.

Participants will be asked to:

* Lie inside an MRI scanner for up to 90 minutes (including breaks), in different body positions
* Undergo NIV therapy for 5-10 minutes while breathing normally inside an MRI scanner
* Have their upper airway resistance measured, in different body positions

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18+
* Willing and able to consent to the study

Exclusion Criteria:

* Contraindications for MRI (such as metal implants)
* Contraindications for NIV (such as pneumothorax)
* No history of lung or upper airway disease
* Claustrophobia
* Symptoms of a cold, flu, or significant congestion, within the last 3 days
* Self-reported confirmed or suspected pregnancy
* Palatal abnormalities or previous upper airway surgery (such as cleft palate and/or UPPP)
* Prior major head or neck surgery with or without irradiation (such as radiotherapy of cutaneous cancers, robotic surgery for an oropharyngeal cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Volumetric change of soft palate airway size in delta millimeters cubed, | Single 2 hour visit
  millimeters cubed

SECONDARY OUTCOMES:
Impact of positive pressure ventilation on airway volume in millimeters cubed, | Single 2 hour visit
  Change in soft palate airway size with addition of positive pressure ventilation, measured from segmented MRI data of soft palatal airway, and expressed in millimeters cubed, and delta millimeters cubed
Upper airway resistance measurements | Single 2 hour visit
  Changes in upper airway resistance based on different body positions, measured using anterior rhinomanometry according to international guidelines and resistance units expressed as Pa/cm3/s

CONTACTS AND LOCATIONS:
Overall Officials: Alys Clark, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- University of Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided
De-identified and anonymized study data may be shared for further statistical analysis